CLINICAL TRIAL: NCT00079144
Title: Treatment Of Patients With Metastatic Melanoma Using Nonmyeloablative But Lymphocyte Depleting Regimen Followed By The Administration Of In Vitro Sensitized Lymphocytes Reactive With ESO-1 Antigen
Brief Title: Lymphocyte-Depleting Nonmyeloablative Preparative Chemotherapy Followed By Autologous Lymphocyte Infusion, Peptide Vaccine Plus Montanide ISA-51, and Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000354491; NCI-04-C-0104; NCI-6233; NCT00076661 (obsolete NCT alias)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2005-05

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Filgrastim; incomplete Freund's adjuvant; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Biological: NY-ESO-1 peptide vaccine
Biological: aldesleukin
Biological: filgrastim
Biological: incomplete Freund's adjuvant
Biological: therapeutic autologous lymphocytes
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide and fludarabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Treating a person's lymphocytes in the laboratory and reinfusing them may replace immune cells destroyed by chemotherapy. Vaccines made from peptides may make the body build an immune response to kill tumor cells. Giving a vaccine with Montanide ISA-51 may cause a stronger immune response and kill more tumor cells. Interleukin-2 may stimulate a person's lymphocytes to kill tumor cells.

PURPOSE: This phase II trial is studying how well lymphocyte-depleting nonmyeloablative (not damaging to bone marrow) chemotherapy followed by autologous lymphocyte infusion, peptide vaccine plus Montanide ISA-51, and interleukin-2 works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical tumor regression in patients with metastatic melanoma treated with a lymphocyte-depleting nonmyeloablative preparative chemotherapy regimen followed by autologous lymphocyte infusion, ESO-1 peptide vaccination comprising ESO-1:157-165 (165V) and Montanide ISA-51, and interleukin-2.

Secondary

* Determine the survival of the infused lymphocytes in patients treated with this regimen.
* Determine the long-term immune status of patients treated with this regimen.

OUTLINE: Patients are stratified according to type of lymphocyte infusion (ESO-1-reactive tumor-infiltrating lymphocytes [TIL] vs ESO-1 reactive peripheral blood lymphocytes [PBL]).

* Autologous lymphocyte collection and expansion: Autologous PBL or TIL are collected from patients during leukapheresis or biopsy. The cells are sensitized in vitro with ESO-1:157-165 (165V) melanoma antigen and expanded.
* Lymphocyte-depleting nonmyeloablative preparative chemotherapy: Patients receive lymphocyte-depleting nonmyeloablative preparative chemotherapy comprising cyclophosphamide IV over 1 hour on days -7 and -6 and fludarabine IV over 15-30 minutes on days -5 to -1.
* Autologous lymphocyte infusion: Autologous PBL or TIL are reinfused on day 0*. Patients also receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 1 and continuing until blood counts recover.
* ESO-1 peptide vaccination: Patients receive ESO-1 peptide vaccination comprising ESO-1:157-165 (165V) peptide emulsified in Montanide ISA-51 SC on days 0*-4, 11, 18, and 25.
* Interleukin therapy: Patients receive interleukin-2 IV over 15 minutes 3 times daily on days 0*-4.

NOTE: *Day 0 is 1-4 days after the last dose of fludarabine.

Patients achieving stable disease or partial response may receive up to 1 retreatment course. Patients with progressive disease after infusion of PBL may receive retreatment with TIL, if available.

Patients are followed at 4-5 weeks, every 3-4 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 24-74 patients (12-37 per stratum) will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma that is refractory to standard therapy (including high-dose interleukin-2)
* Measurable disease
* HLA-A*0201 positive
* Epstein-Barr virus positive
* ESO-1-expressing disease by reverse transcription polymerase chain reaction amplified tissue OR presence of ESO-1 serum antibody

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 8.0 g/dL

Hepatic

* Hepatitis B surface antigen negative
* Hepatitis C antibody negative
* AST and ALT < 3 times upper limit of normal
* Bilirubin ≤ 2.0 mg/dL (< 3.0 mg/dL for patients with Gilbert's syndrome)
* No coagulation disorders

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No prior myocardial infarction
* No major cardiovascular illness by stress thallium or comparable test
* No cardiac arrhythmias
* LVEF ≥ 45%
* Normal cardiac stress test required for the following conditions:

  * Prior EKG abnormalities
  * Symptoms of cardiac ischemia
  * Arrhythmias
  * Age 50 and over

Pulmonary

* FEV_1 > 60% of predicted (for patients with a prolonged history of cigarette smoking or symptoms of respiratory dysfunction)
* No obstructive or restrictive pulmonary disease
* No other major respiratory illness

Immunologic

* HIV negative
* No active systemic infection
* No opportunistic infection
* No major immune system illness
* No form of primary or secondary immunodeficiency
* No known hypersensitivity to study agents

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 4 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* Prior ESO-1-based vaccination allowed

Chemotherapy

* At least 6 weeks since prior nitrosoureas and recovered

Endocrine therapy

* No concurrent systemic steroid therapy

Radiotherapy

* Recovered from prior radiotherapy

Surgery

* Not specified

Other

* At least 4 weeks since prior systemic therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-01; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Clinical tumor regression

SECONDARY OUTCOMES:
Survival of infused lymphocytes
Long-term immune status

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland